CLINICAL TRIAL: NCT01395381
Title: Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Benefit of Antihelminthic Therapy in the Community-Based Treatment of Severe Acute Malnutrition in Malawian Children
Brief Title: Effectiveness of Oral Albendazole in the Treatment of Severe Acute Malnutrition
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not funded
Sponsor: Washington University School of Medicine (Other)
Collaborators: Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MJM-albendazole
Record Dates: First submitted 2011-07-01; First posted 2011-07-15 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Kwashiorkor; Marasmus
MeSH Terms: conditions — Kwashiorkor; Protein-Energy Malnutrition | interventions — Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Albendazole (Experimental)
  Interventions: Drug: Albendazole

INTERVENTIONS:
Drug: Placebo — placebo given once
  Arms: Placebo
Drug: Albendazole — single dose albendazole given at the time of enrollment
  Arms: Albendazole

SUMMARY:
The benefit of anti-worm therapy as part of the case management of severe acute malnutrition (SAM) in the outpatient setting has not previously been studied. This study will compare recovery rates of children with SAM treated in the community with locally-produced ready-to-use therapeutic food (RUTF) with and without prescribed albendazole as part of their case management.

ELIGIBILITY:
Inclusion Criteria:

* 12-59 months old
* Kwashiorkor and/or Marasmus
* Qualified for home-based therapeutic feeding with RUTF

Exclusion Criteria:

* Obvious congenital or other malformation that makes child a poor candidate for feeding with RUTF
* Unable to consume test-dose of RUTF in clinic
* Parent refusal to participate and return for follow-up

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
nutritional recovery | 12 weeks
  Weight-for-Height Z-score (WHZ) > -2 without bipedal pitting edema
mortality | 12 weeks

SECONDARY OUTCOMES:
malnutrition relapse | 6 months
  acute malnutrition, either moderate (WHZ < -2) or severe (WHZ < -3 and/or bipedal pitting edema)
height and weight gain | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, MD, Principal Investigator — University of Malawi; Kenneth Maleta, MBBS PhD, Principal Investigator — University of Malawi; Indi Trehan, MD MPH DTM&H, Study Director — University of Malawi
Locations (1):
- St. Louis Nutrition Project, Blantyre, Malawi